CLINICAL TRIAL: NCT07400471
Title: The Effects of Preemptive Multimodal Analgesic on Endodontic Pain.
Brief Title: The Effects of Preemptive Multimodal Analgesic on Endodontic Pain Following Root Canal Therapy.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chattogram International Dental College (Other)
Responsible Party: Principal Investigator, Prof. Dr. Md. Abu Saeed Ibn Harun, Professor, Chattogram International Dental College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ERC-BBS/2025/0015-44/2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post Endodontic Pain; Mechanical Detection Threshold; Mechanical Pain Threshold; Mechanical Pain Sensitivity
Keywords: post endodontic pain; Root canal Therapy; Multimodal Analgesia; Dynamic sensory test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Consequently, triple binding is ensured (by the sit investigator, patient, and operator). The statistician in charge of the data analysis will also be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Analgesia (Active Comparator): Preemptive Multi modal analgesic drug: Experimental group will be divided into 2 subgroups according to use of drug.
  A. Pregabalin-acetaminophen. B. Duloxetine-Acetaminophen Pregabalin-acetaminophen: Before a half-hour endodontic treatment, patients in this group will receive a single dosage of 50 mg pregabalin and 500 mg acetaminophen. If necessary, acetaminophen dosages of 500 mg will be administered three times a day.
  Duloxetine-Acetaminophen: Prior to a half-hour endodontic treatment, patients in this group will receive a single dosage of 500 mg of acetaminophen and 30 mg of Duloxetine. If necessary, acetaminophen dosages of 500 mg will be administered three times a day.
  Interventions: Drug: Pregabalin- Acetaminophen; Drug: Duloxetine- Acetaminophen
- Control (Placebo Comparator): Placebo: Patient in this group will receive placebo drug before half an hour of operating procedure. If necessary, acetaminophen dosages of 500 mg will be administered three times a day and noted
  Interventions: Drug: Pregabalin- Acetaminophen; Drug: Duloxetine- Acetaminophen

INTERVENTIONS:
Drug: Pregabalin- Acetaminophen — Preemptive Multi modal analgesic drug: Experimental group will be divided into 2 subgroups according to use of drug.
  A. Pregabalin-acetaminophen. B. Duloxetine-Acetaminophen Pregabalin-acetaminophen: Before a half-hour endodontic treatment, patients in this group will receive a single dosage of 50 mg pregabalin and 500 mg acetaminophen. If necessary, acetaminophen dosages of 500 mg will be administered three times a day.
Drug: Duloxetine- Acetaminophen — Duloxetine-Acetaminophen: Prior to a half-hour endodontic treatment, patients in this group will receive a single dosage of 500 mg of acetaminophen and 30 mg of Duloxetine. If necessary, acetaminophen dosages of 500 mg will be administered three times a day.

SUMMARY:
A clinical trial comparing preemptive multimodal analgesics with placebo in the management of immediate and chronic post-endodontic pain. The study utilizes statistical methods such as chi-squared, T-tests, and regression analysis, accounting for multiple outcomes with the Bonferroni adjustment. Duloxetine hydrochloride and pregabalin, both available in Bangladesh, are evaluated as experimental drugs, while placebos are used to assess psychological effects on pain. All participants receive standard interventional treatments, with acetaminophen provided as needed, and ethical considerations are addressed according to international guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's aged 18 years more.
2. ASA physical status I-II.
3. Patient with the complain of pain originated from teeth and surrounding structure.
4. Preoperative pain severity is moderate to severe.
5. Patient can be able to make communication about their pain.
6. Patients give consent to attain this research.
7. Patients have others concomitant chronic pain.
8. Patients who will have non-surgical endodontic treatment.
9. Patients who will have non-surgical endodontic retreatment.
10. Patients who will have surgical endodontic treatment.

Exclusion Criteria:

1. Patient would not like to attain in research.
2. Patients have any medical condition those are contra indication for study drug.
3. ASA physical status III, IV, V.
4. Patient already under treated any anti convulsent drug.
5. Patient participant in other clinical trials.
6. Lack of motivation or poor adharence to study protocols.
7. Patient with Pregnancy
8. Severe organ dysfunction
9. Patient have Hepatitis B, and other cross infection disease like (HIV)
10. Uncontrolled comorbidities that patient do not fit for endodontic treatment.
11. Severe cognitive impaired patients.
12. History of certain cancers or severe hematological issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Effects of Preemptive multimodal analgesia on post endodontic pain | 6, 12, 24, 48, 72 hours
  Primary Pain during endodontic treatment and the effectiveness of intervention will be evaluated at 6, 12, 24, 48, 72, and hourly intervals after the endodontic procedure. Treatment-related anaesthetic efficacy will be assessed using the VAS (Visual Analogue Scale; numerical value 0-10). During endodontic treatment, the level of pain will decide how effective the anesthetic is. The patient will be asked to rate the analgesic effects on a VAS (Visual Analogue Scale) scale by providing a numerical number 0-10. '0" are indicated no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= sever pain.

SECONDARY OUTCOMES:
Mechanical Detection Threshold | baseline, 72 hours
  Mechanical Detection Threshold: A standardized set of modified von Frey hairs (Opti-hair2-Set, Marstock Nervtest, Germany) that exert stresses upon bending between 0.25 and 512 mN graded by a factor of 2 (1-2 s contact time) were used to determine the mechanical detection threshold (MDT). With a rounded tip and 0.5 mm in diameter, the von Frey hairs' contact area with the skin was consistent in size and shape to prevent sharp edges that could aid in nociceptor activation. Five threshold determinations with a sequence of increasing and decreasing stimulus intensities were made using the "method of limits." The geometric mean of these five series served as the final threshold.
Mechanical Pain Threshold | baseline, 72 hours
  Mechanical Pain Threshold: A set of seven pin-prick mechanical stimulators with preset stimulus intensities (flat contact area of 0.2 mm diameter) that applied forces of 8, 16, 32, 64, 128, 256, and 512 mN were used to test the mechanical pain threshold (MPT). These stimuli were custom-made and weighted. Until the first perception of sharpness was attained, the stimulators were applied in ascending order at a pace of two seconds on, two seconds off. The geometric mean of five sequences of rising and descending stimuli served as the final threshold. The purpose of this test was to identify pinprick hypoalgesia. Before initiation of endodontic treatment, the patient has to take drug that's are supplied in enveloped.
Mechanical Pain Sensitivity | baseline, 72 hours
  Mechanical Pain Sensitivity will test using the same weighted pinprick stimuli as for mechanical pain threshold. To obtain a stimulus- response- function, these seven pinprick stimuli will apply in a balanced order, five times each, and patient will ask to give a pain rating for each stimulus on a 0-10 VAS scale ( '0' indicate no pain; 10 indicate most intense pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Professor. Dr. Md. Abu Saeed Ibn Harun, Chittagong, Chattogram, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anibal Diogenes, Michael A. Henry. Pain Pathways and Mechanisms of the Pulpodentin Complex. Chapter 8; Seltzer and Bender's Dental Pulp. 2nd edition. Quintessence Publishing Co Inc;2012.
- [Background] Jang YE, Kim Y, Kim BS. Influence of Preoperative Mechanical Allodynia on Predicting Postoperative Pain after Root Canal Treatment: A Prospective Clinical Study. J Endod. 2021 May;47(5):770-778.e1. doi: 10.1016/j.joen.2021.01.004. Epub 2021 Jan 29. PMID 33516824
- [Background] Alelyani AA, Azar PS, Khan AA, Chrepa V, Diogenes A. Quantitative Assessment of Mechanical Allodynia and Central Sensitization in Endodontic Patients. J Endod. 2020 Dec;46(12):1841-1848. doi: 10.1016/j.joen.2020.09.006. Epub 2020 Sep 15. PMID 32941893
- [Background] Wiech K, Ploner M, Tracey I. Neurocognitive aspects of pain perception. Trends Cogn Sci. 2008 Aug;12(8):306-13. doi: 10.1016/j.tics.2008.05.005. Epub 2008 Jul 5. PMID 18606561
- [Background] Md. Abu Saeed Ibn Harun et al. The dimension and severity of orofacial pain in patients with current and chronic odontogenic pain. M Dent J 2021; 41(3): 235-244.
- [Background] Woolf CJ. Windup and central sensitization are not equivalent. Pain. 1996 Aug;66(2-3):105-8. No abstract available. PMID 8880830
- [Background] Md. Abu Saeed Ibn Harun et al. Endogenous Pain modulation of Irreversible Pulpitis and Persistent Endodontic Pain. Chattagram International Dental College Journal 2019; 2(1):9-13.
- [Background] O'Keefe EM. Pain in endodontic therapy: preliminary study. J Endod. 1976 Oct;2(10):315-9. doi: 10.1016/S0099-2399(76)80047-7. No abstract available. PMID 1068208
- [Background] Doleman B, Leonardi-Bee J, Heinink TP, Boyd-Carson H, Carrick L, Mandalia R, Lund JN, Williams JP. Pre-emptive and preventive NSAIDs for postoperative pain in adults undergoing all types of surgery. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD012978. doi: 10.1002/14651858.CD012978.pub2. PMID 34125958
- [Background] Price DD, Finniss DG, Benedetti F. A comprehensive review of the placebo effect: recent advances and current thought. Annu Rev Psychol. 2008;59:565-90. doi: 10.1146/annurev.psych.59.113006.095941. PMID 17550344
- [Result] Ince B, Ercan E, Dalli M, Dulgergil CT, Zorba YO, Colak H. Incidence of postoperative pain after single- and multi-visit endodontic treatment in teeth with vital and non-vital pulp. Eur J Dent. 2009 Oct;3(4):273-9. PMID 19826598
- [Result] Al-Nahlawi T, Alabdullah A, Othman A, Sukkar R, Doumani M. Postendodontic pain in asymptomatic necrotic teeth prepared with different rotary instrumentation techniques. J Family Med Prim Care. 2020 Jul 30;9(7):3474-3479. doi: 10.4103/jfmpc.jfmpc_342_20. eCollection 2020 Jul. PMID 33102316
- [Result] Nixdorf DR, Moana-Filho EJ, Law AS, McGuire LA, Hodges JS, John MT. Frequency of persistent tooth pain after root canal therapy: a systematic review and meta-analysis. J Endod. 2010 Feb;36(2):224-30. doi: 10.1016/j.joen.2009.11.007. PMID 20113779
- [Result] Oshima K, Ishii T, Ogura Y, Aoyama Y, Katsuumi I. Clinical investigation of patients who develop neuropathic tooth pain after endodontic procedures. J Endod. 2009 Jul;35(7):958-61. doi: 10.1016/j.joen.2009.04.017. PMID 19567314
- [Result] Hargreaves KM, BermanLH, Cohen S. Cohen's Pathways of the Pulp. 11th ed. Amsterdam, Netherlands: Elsevier; 2015.
- [Result] Santos-Puerta N, Penacoba-Puente C. Pain and Avoidance during and after Endodontic Therapy: The Role of Pain Anticipation and Self-Efficacy. Int J Environ Res Public Health. 2022 Jan 27;19(3):1399. doi: 10.3390/ijerph19031399. PMID 35162422
- [Result] Smith EA, Marshall JG, Selph SS, Barker DR, Sedgley CM. Nonsteroidal Anti-inflammatory Drugs for Managing Postoperative Endodontic Pain in Patients Who Present with Preoperative Pain: A Systematic Review and Meta-analysis. J Endod. 2017 Jan;43(1):7-15. doi: 10.1016/j.joen.2016.09.010. Epub 2016 Dec 6. PMID 27939729
- [Result] Suneelkumar C, Subha A, Gogala D. Effect of Preoperative Corticosteroids in Patients with Symptomatic Pulpitis on Postoperative Pain after Single-visit Root Canal Treatment: A Systematic Review and Meta-analysis. J Endod. 2018 Sep;44(9):1347-1354. doi: 10.1016/j.joen.2018.05.015. Epub 2018 Jul 24. PMID 30054100
- [Result] Zanjir M, Sgro A, Lighvan NL, Yarascavitch C, Shah PS, da Costa BR, Azarpazhooh A. Efficacy and Safety of Postoperative Medications in Reducing Pain after Nonsurgical Endodontic Treatment: A Systematic Review and Network Meta-analysis. J Endod. 2020 Oct;46(10):1387-1402.e4. doi: 10.1016/j.joen.2020.07.002. Epub 2020 Jul 12. PMID 32668310
- [Result] Mazaleuskaya LL, Theken KN, Gong L, Thorn CF, FitzGerald GA, Altman RB, Klein TE. PharmGKB summary: ibuprofen pathways. Pharmacogenet Genomics. 2015 Feb;25(2):96-106. doi: 10.1097/FPC.0000000000000113. No abstract available. PMID 25502615
- [Result] Compound Summery Acetaminophen. National Library of Medicine. Seen 2023. www.pubchem.ncbi.nlm.nih.gov.
- [Result] Park SJ, Zhang S, Chiang CY, Hu JW, Dostrovsky JO, Sessle BJ. Central sensitization induced in thalamic nociceptive neurons by tooth pulp stimulation is dependent on the functional integrity of trigeminal brainstem subnucleus caudalis but not subnucleus oralis. Brain Res. 2006 Sep 27;1112(1):134-45. doi: 10.1016/j.brainres.2006.06.115. Epub 2006 Aug 22. PMID 16930568
- [Result] 37. Harun, A. S. I. harun, Hossain, . A., Jabber, S. and Hasan, H. . (2021) "The dimension and severity of orofacial pain in patients with current and chronic odontogenic pain", Mahidol Dental Journal. Bangkok, Thailand, 41(3), pp. 235-244. available at: https://he02.tci-thaijo.org/index.php/mdentjournal/article/view/251124 (accessed: 3 June 2025).